CLINICAL TRIAL: NCT02497794
Title: Efficacy and Effectiveness of Gum Chewing on Bowel Function After Cesarean Section: a Randomized Controlled Trial
Brief Title: The Effect of Gum Chewing on Bowel Function After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nazlı YENIGUL, doctor, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 787
Record Dates: First submitted 2015-06-28; First posted 2015-07-15 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Splinter of Gum
Keywords: chew gum; bowel movements; cesarean section
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- postoperative chew gum (Active Comparator): The patients in the study group will chew one sugarless gum for 30 minutes in postoperative 3., 5. and 7. hours.
  Interventions: Other: chew gum
- without postoperative chew gum (Placebo Comparator): The control group will be followed without chew gum.
  Interventions: Other: chew gum

INTERVENTIONS:
Other: chew gum — The patients in the study group,will chew one sugarless gum for 30 minutes in postoperative 3., 5. and 7. hours. The control group will be followed without chew gum. Both patient groups will be mobilized in postoperative 6 hour and 8 hour after the operation, juicy food will be given. It will be introduced to solid foods after bowel movements and gas output occurs. All patients postoperatively 4, 6,8,10., 12., 24 and 48 hours will be examined and bowel sounds will be oscult. Gas evolution is still not, enema will be applied. All patients will note the time of first rumbling of the stomach, first feeling of hunger and the first gas outlet.
  Other Names: postoperative chew gum

SUMMARY:
This study is a randomised controlled trial that included 150 pregnant women undergoing cesarean in Sisli Ethal Training and Research Hospital, Department of Obstetrics and Gynecology, Istanbul, Turkey. It was carried out in the period from October 1, 2015 to December 31, 2015. After operation, the participants are going to randomly assigned into two groups by using cards. The patients are going to randomized into two groups by using a sealed enveloped system.The patients in the study group, will chew one sugar less gum for 30 minutes in postoperative 3., 5. and 7. hours. The control group will be followed without chew gum. All patients will note the time of first rumbling of the stomach, first feeling of hunger and the first gas outlet.

DETAILED DESCRIPTION:
For elective cases, all participants are going to given nothing by mouth since midnight before surgery, and all operations are going to perform in the morning. For those who had emergency cesarean section, nothing is going to given per oral for at least 4 hours before the start of the operation. Operation data is going to recorded including surgical setting, type of cesarean section, previous surgery, adhesion and operation time.

After operation, the participants are going to randomly assigned into two groups by using cards. The patients are going to randomized into two groups by using a sealed enveloped system. A blue card and an orange card are going to sealed in separate envelopes. Blue card means patients will chewgum.

The patients in the study group, will chew one sugar less gum for 30 minutes in postoperative 3., 5. and 7. hours. The control group will be followed without chew gum. Both patient groups will be mobilized in postoperative 6 hour and 8 hour after the operation, juicy food will be given. It will be introduced to solid foods after bowel movements and gas output occurs. All patients postoperatively 4, 6, 8, 10, 12, 24 and 48 hours will be examined and bowel sounds will be oscult. Gas evolution is still not, enema will be applied. All patients will note the time of first rumbling of the stomach, first feeling of hunger and the first gas outlet.

ELIGIBILITY:
Inclusion Criteria:

1. pregnant women who is at least 18 years of age
2. pregnant women whose body mass index is under 35
3. pregnant women who is going to have cesarean section.

Exclusion Criteria:

1. cesarean hysterectomy,
2. surgical management of severe postpartum hemorrhage
3. previous bowel surgery
4. women with history of drug consumption,especially opioids
5. water and electrolyte disturbances
6. pancreatitis or peritonitis
7. inability to chew gum
8. diabetes, pregnancies accompanied by coagulopathy like pre-eclampsia, hypothyroidism, muscular and neurological disorders
9. postoperative admission to intensive care unit
10. history of abdominal surgery except cesarean section
11. history of postoperative ileus
12. patients with drains

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Postoperative time to return to active bowel movements | up to 48 hours
  The investigators are going to examine all patients postoperatively 4, 6,8,10., 12., 24 and 48 hours and oscult the bowel sounds. Also all patients are going to note the time of first rumbling of the stomach, first feeling of hunger and the first gas outlet.

SECONDARY OUTCOMES:
Postoperative infection rates and early discharge | up to 48 hours
  Postoperative ileus and general surgery consultation were recorded. After discharge, all patients were called post-op sixth day control.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma YAZICI YILMAZ, Principal Investigator — Sisli etfal; Begüm AYDOGAN, Study Director — Sisli etfal
Locations (1):
- Sisli Etfal Research and Training hospital, Obstetrics and gynecology department, Istanbul, Marmara, Turkey (Türkiye)